CLINICAL TRIAL: NCT07042607
Title: The Role of Dysfunctional Schemas and Acceptance Regarding Chronic Fatigue in Oncology Patients After Treatment
Acronym: CVONCOS
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Marianne van der Zijden, drs, Zuyderland Medisch Centrum
Other Study IDs: METCZ20220084
Record Dates: First submitted 2024-08-19; First posted 2025-06-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Fatigue
Keywords: dysfunctional schema; acceptance; chronic fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- not appicable: not appicable
  Interventions: Other: not appicable

INTERVENTIONS:
Other: not appicable — no intervention

SUMMARY:
The role of dysfunctional schemas and acceptance regarding chronic fatigue in oncology patients after treatment

This scientific cross-sectional study is at the intersection of medical psychology and oncology and will address the role of dysfunctional schemas and acceptance in the development of fatigue symptoms after treatment for cancer.

DETAILED DESCRIPTION:
Cancer is potentially a deadly disease, but early detection and modern available treatments have increased survival rates in recent decades. Increasing attention is being paid to the well-being of survivors. One of the side effects of long-term curative treatment of cancer, is chronic fatigue. Fatigue has a major impact on daily life and thus on the patient's quality of life.

This study deals with patients who still suffer from chronic fatigue 6 months to two years after (intentionally curative) cancer treatment. Defined in English as chronic cancer-related fatigue (CCRF). The role of acceptance and dysfunctional schedules in maintaining chronic fatigue after cancer will be investigated.

The question is whether oncology patients with dysfunctional schedules after treatment are more likely to maintain CCRF than oncology patients in whom these dysfunctional schedules are present to a lesser extent. From the literature, we chose to examine the dysfunctional schema Relentlessly strict standards/extremely high demands. Exploratively, we also examine the dysfunctional schemas Abandonment/Instability and Self-Sacrifice.

If the above schemas are indeed associated with higher levels of CCRF, we then ask what role acceptance of fatigue plays on the aforementioned correlation. We hypothesize that acceptance plays a mediating role in the correlation between dysfunctional schemas and fatigue: Dysfunctional schemas hinder acceptance of fatigue. Next, we hypothesize that the lower the degree of acceptance, the higher the perceived fatigue will be.

In addition to mediation, a moderating role of dysfunctional schemas could also be hypothesized. Therefore, the second hypothesis hypothesizes that there is a negative relationship between acceptance and fatigue, but only when the relevant dysfunctional schemas are present at low levels. When these dysfunctional schemas are present to a high degree, the relationship between acceptance and fatigue changes. Most likely, the dysfunctional schemas reduce the beneficial influence of acceptance.

ELIGIBILITY:
Inclusion Criteria:

* All oncology patients (18 up to and including 70 years of age ), at least 6 months to no later than five years after the last curative treatment and have had no other oncology treatment thereafter (except hormone therapy). The type of oncology treatment (chemotherapy, radiotherapy, immunotherapy or hormone therapy) and the type of cancer they have had are diverse. Subjects recruited should have a good command of the Dutch language in connection with optimal reading and answering of the questionnaires.

Exclusion Criteria:

Exclusion criteria for participation are a psychotic disorder and current substance dependence.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All oncology patients (18 up to and including 70 years of age), at least 6 months to no later than five years after the last curative treatment and have had no other oncology treatment thereafter (except hormone therapy)
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Fatigue | Baseline
  The Individual Stress Strength Checklist measures subjective fatigue and behavioral aspects related to it. It consists of 20 statements that examine how the respondent has felt over the past two weeks, indicating to what extent the statement applies to him/her. It measures a picture of fatigue that includes fluctuations over time. Four subscales are distinguished. The scoring method is on a 7-point Likert scale. A cut-off point for the total score is 76, indicating problematic fatigue. For the subjective fatigue subcategory, Normal = a score below 27. A score of 27 or higher is an indication of abnormal fatigue. A score of 35 or higher is considered an indication of severe fatigue.
Dysfunctional schema | Baseline
  The Young Schema Questionnaire-S3 (YSQ-S3) provides insight into dysfunctional schemas that may be underlying patients' psychological problems. The YSQ-S3 consists of 90 items (statements) measuring 18 schemas including the dysfunctional schemas of ruthless standards/excessive demands, self-sacrifice and abandonment. The method of scoring is on a 6-point Likert scale. After taking the YSQ-S3, the average of all scores per scale is calculated for high predictive value. For most schema scales, a mean score of 2.5 or higher usually appears to fall in the clinical range. The cut-off value for Self-sacrifice and Compassionate norms/extreme demands is around a mean of 3. Internal consistency is adequate for all 18 scales: Cronbach's α=0.70
Acceptance | Baseline
  The Freiburg mindfulness Inventory-Short Form (FMI-SF) is a questionnaire consisting of two subscales: Presence (attention to experiences of the present moment) and Acceptance (an accepting attitude toward experiences). The FMI-SF has the advantage of being a short list of 14 questions that can be applied in a clinical setting. The items can be scored from 1 (rarely) to 4 (almost always). Both the FMI-14 as a whole (Cronbach's α = .85) and the factors Presence (Cronbach's α= .74) have adequate internal consistency, providing support for the reliability of the scale and subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Marianne van der Zijden, Heerlen, Limburg, Netherlands